CLINICAL TRIAL: NCT00005097
Title: A Randomized, Double-Blind, Placebo-Controlled Phase II Clinical Trial of Polyphenon E Against Various Endpoints of Actinic Keratosis Pathobiology
Brief Title: Green Tea Extract in Treating Patients With Actinic Keratosis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: terminated due to the low conditional power for a positive study
Sponsor: Frank Meyskens (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Frank Meyskens, Cancer Center, University of California, Irvine
Organization: University of California, Irvine (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: UCI 98-31 / CDR0000067798; UCIRVINE-N01-CN-85182 (Other: UC Irvine); NCI-P00-0142 (Registry Identifier: National Cancer Insitute); UCI 98-31 (Other: University of California, Irvine); 1998-420 (Other: University of California, Irvine)
Record Dates: First submitted 2000-04-06; First posted 2004-04-02 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Non-melanomatous Skin Cancer
Keywords: squamous cell carcinoma of the skin
MeSH Terms: interventions — polyphenon E

STUDY DESIGN:
Intervention Model Description: Subjects will have actinic keratosis on both arms and apply Polyphenon E topical ointment on one arm and placebo ointment to apply to the other arm. Subjects will serve as their own control by being unaware of which arm will have the active study drug.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Polyphenon E & Placebo (Experimental): Each subject will receive both the Polyphenon E and placebo, one on each arm.
  One arm will be assigned to be treated with topical Polyphenon E daily for 12 weeks and the other with placebo vehicle in a random, double blind manner daily for 12 weeks.
  Interventions: Drug: Polyphenon E and Placebo

INTERVENTIONS:
Drug: Polyphenon E and Placebo — Areas of sun damaged skin with actinic keratoses to be treated will be mapped and photographed on patient's bilateral arms. One of the patient's arms will be assigned to be treated with topical Polyphenon E, the patient's other arm with placebo vehicle in a random, double blind manner. The patient's arm treatment areas will receive daily applications of a premeasured amount of drug or placebo. Patients will be seen every other week for 12 weeks to check for effects of the applications and monitor for compliance or possible side effects.
  Other Names: kunecatechins ointment and placebo

SUMMARY:
RATIONALE: Green tea extract contains ingredients that may inhibit the growth of actinic keratosis.

PURPOSE: Randomized phase II trial to determine the effectiveness of green tea extract in treating patients who have actinic keratosis.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the efficacy of the green tea extract epigallocatechin gallate (Polyphenon E topical ointment) in causing complete clinical and histopathologic regression in patients with actinic keratoses. II. Determine duration of treatment with Polyphenon E necessary to cause regression in these patients. III. Describe pathophysiologic and molecular alterations in actinic keratoses and sun damaged skin that are not present in skin that is not sun damaged in these patients. IV. Determine the effects of this treatment on biomarkers for skin cancer in these patients.

OUTLINE: This is a randomized, double blind, placebo controlled study. One of the patient's arms is randomized to receive topical epigallocatechin gallate (Polyphenon E), the other arm to receive a placebo. Patients receive topical applications daily for 12 weeks, or until resolution of all actinic keratoses within the treatment field.

PROJECTED ACCRUAL: A minimum of 60 patients will be accrued for this study over 10 months.

ELIGIBILITY:
Inclusion Criteria:

1. participants multiple sites of actinic keratosis identified by clinical examination and the histologic confirmation of one lesion (Grade 1-3 as defined previously in "Clinical Grading") are eligible.
2. No history of invasive cancer within 5 years (though non-melanoma skin cancer, stage I cervical cancer, or chronic lymphocytic leukemia (CLL) stage 0 will not be reason to exclude a patient); no severe metabolic disorders or other life-threatening acute or chronic disease; no additional x-ray or chemotherapy anticipated.
3. Not requiring use of topical medications in areas being studied.
4. Subjects must meet the Southwest Oncology Group performance status criteria of 0 - 1 (0= fully active, able to carry on all pre-disease activities without restriction [Karnofsky scale 90 - 100]; 1 = restricted in physically strenuous activity, but ambulatory and able to carry out work of a light or sedentary nature, i.e. light housework or office work [Karnofsky scale 70 - 80]).
5. Signed informed consent approved by the local Human Subjects Committee (Institutional Review Board).

Exclusion Criteria:

1. Use of the following systemic or local therapies for the periods specified, prior to entry into the study:

   Within 2 weeks: topical medications, e.g. corticosteroids, alpha-hydroxyacids (glycolic acid, lactic acid) or retinoids (Retin-A) to the target lesions Within 4 weeks: systemic steroid therapy. Within 2 months: cryotherapy to the target lesions, laser resurfacing, chemical peels, topical application of 5-fluorouracil (5-FU) or masoprocol (Actinex) for treatment of actinic keratoses. Systemic treatment with chemotherapeutic agents, psoralens, immunotherapy, retinoids (Tegison, Accutane).
2. Any medical condition which , in the opinion of the investigator, could preclude study participation
3. Active infectious diseases such as tuberculosis (TB) or HIV that may affect the patient systemically and may also affect the immune system. Localized, minor infections such as sinusitis, uncomplicated urinary tract infection, otitis media, etc. will not be criteria for exclusion from the study.
4. Use of any investigational drug in the previous 30 days.
5. Any history of keloid formation.
6. Pregnant or nursing patients.
7. Participants who may be unreliable for the study, including those engaging in excessive alcohol intake or drug abuse, or participants who are unable to return for scheduled follow-up visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 1999-08; Primary Completion 2002-08 (Actual); Study Completion 2002-08 (Actual)

PRIMARY OUTCOMES:
Clinical and histopathologic regression of actinic keratoses | 12 weeks
  Measure efficacy of Polyphenon E in causing complete and clinical and histopathologic regression of actinic keratoses in comparison to placebo

CONTACTS AND LOCATIONS:
Overall Officials: Frank L. Meyskens, MD, FACP, Study Chair — Chao Family Comprehensive Cancer Center
Locations (1):
- Chao Family Comprehensive Cancer Center, Orange, California, United States

REFERENCES:
- [Result] Carpenter PM, Linden KG, McLaren CE, Li KT, Arain S, Barr RJ, Hite P, Sun JD, Meyskens FL Jr. Nuclear morphometry and molecular biomarkers of actinic keratosis, sun-damaged, and nonexposed skin. Cancer Epidemiol Biomarkers Prev. 2004 Dec;13(12):1996-2002. PMID 15598753
- [Result] Linden KG, Carpenter PM, McLaren CE, Barr RJ, Hite P, Sun JD, Li KT, Viner JL, Meyskens FL. Chemoprevention of nonmelanoma skin cancer: experience with a polyphenol from green tea. Recent Results Cancer Res. 2003;163:165-71; discussion 264-6. doi: 10.1007/978-3-642-55647-0_15. PMID 12903852